CLINICAL TRIAL: NCT05222373
Title: Community-based Cognitive Behavioral Lifestyle Therapy to Improve Diabetes-Related Health Outcomes in an Underserved Latino Population
Brief Title: Community-based CBT and T2D in Latino Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Collaboration with partner organization ended.
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Julia López, Assistant Professor in Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202110125; P30DK056341 (NIH)
Record Dates: First submitted 2021-12-22; First posted 2022-02-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes; Mental Health Issue; Quality of Life; Weight Loss
Keywords: Community health worker; Latinx/Hispanic; Mental health; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Weight Loss; Psychological Well-Being; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (No Intervention): Standard care: will include the CHW curriculum focused on diabetes education and connecting individuals to appropriate resources in the community (materials in Spanish and English).
- CBT-based lifestyle intervention group (Active Comparator): CBT-based lifestyle intervention: standard care plus a theoretically-based, diet, activity, and mental health lifestyle intervention integrated within a culturally sensitive curriculum (materials in Spanish and English).
  Interventions: Behavioral: CBT-based lifestyle intervention

INTERVENTIONS:
Behavioral: CBT-based lifestyle intervention — The standard care plus a theoretically-based, diet, activity, and mental health lifestyle intervention integrated within a culturally sensitive curriculum (materials in Spanish and English). Trained CHWs will promote CBT-based lifestyle-change aims and assist in goal setting with participants to reach the primary goal of appropriate glycemic control (fasting blood glucose and HbA1c) and weight reduction, in addition to decrease in depressive symptoms and stress and an increase in quality of life. Participants' body weight, body composition, metabolic measures, and mental health outcomes will be obtained at enrollment and at the end of the intervention.
  Arms: CBT-based lifestyle intervention group

SUMMARY:
The purpose of this project is to develop and test the acceptance and clinical efficacy of a cognitive behavioral therapy (CBT)-based lifestyle intervention, to help manage obesity and diabetes-related health outcomes, provided through community health workers (CHWs) in Latino adults with type 2 diabetes (T2D). A collaboration with an established community-based organization named Sansum Diabetes Research Institute (SDRI), will provide an opportunity to develop, train and implement a culturally sensitive curricula for the CHWs that focuses on body weight and mental health (depressive symptoms and stress) among participants disproportionately impacted by T2D due to social, economic and community factors. Cultural sensitivity focuses on delivering health information based on norms, values, beliefs, environmental factors, and historical context that is unique to a racial/ethnic population. Therefore, for our curricula to be culturally sensitive it will include the following aspects: being primarily delivered in the Spanish language with English as needed, actively incorporate culturally relevant eating and physical activity recommendations, and encompass the foundational importance of familial and social relationships as part of the mental health component of the intervention. For this proposal, the specific aims of this project are: 1) develop a CBT-based lifestyle intervention that focuses on diet, activity, depressive symptoms, stress, and quality of life in collaboration with CHWs and participants from SDRI, and provide training for three CHWs to implement this intervention; 2) conduct a 26-week randomized controlled trial in 50 Latino adults with T2D in the SDRI organization to evaluate the efficacy of the CBT-based lifestyle intervention to improve weight- and diabetes- related health outcomes (body weight, glycemic control, blood pressure, lipid profile, depressive symptoms, stress, and quality of life); 3) evaluate the acceptance and delivery of the CBT-based lifestyle intervention in CHWs and participants with T2D. If successful, this study will establish the structure and content of a culturally sensitive, effective CBT-lifestyle, community-based treatment.

DETAILED DESCRIPTION:
We will implement a CBT-based lifestyle intervention program, among Latino adults with T2D, that targets appropriate body weight, glycemic control, blood pressure, plasma triglyceride, and emphasizes techniques to help reduce depressive symptoms, stress, and improve quality of life through the collaborative partnership with SDRI. Latino adults with T2D who meet eligibility requirements will be recruited for the study, and subjects will be randomized to one of two conditions: 1) Standard care: will include the SDRI CHW curriculum focused on diabetes education and connecting individuals to appropriate resources in the community; or 2) CBT-based lifestyle intervention: standard care plus a theoretically-based, diet, activity, and mental health lifestyle intervention integrated within a culturally sensitive curriculum (materials in Spanish and English).

Trained CHWs will promote CBT-based lifestyle-change aims and assist in goal setting with participants to reach the primary goal of appropriate glycemic control (fasting blood glucose and HbA1c) and weight reduction, in addition to decrease in depressive symptoms and stress and an increase in quality of life. Participants' body weight, body composition, metabolic measures, and mental health outcomes will be obtained at enrollment and at the end of the intervention (week 26).

ELIGIBILITY:
Inclusion Criteria:

i) HbA1c ≥ 6.5% and ≤ 10% at screening; ii) 35 to 65 years old; iii) self-reported Hispanic and/or Latino/a/x heritage; iv) Able to speak and read Spanish; v) obese, defined as BMI 27.0 kg/m2 to 45.0 kg/m2; vi) no change in medications for the past three months; and vii) stable weight (defined as <4% change in body weight) for the past two months.

Exclusion Criteria:

i) treatment with basal insulin >0.5units/kg/day; ii) treatment with rapid acting (prandial) insulin iii) Type 1 diabetes; iv) severe cardiovascular disease defined as: previous stroke, decompensated heart failure New York Heart Association class III or IV, myocardial infarction, unstable angina pectoris, or coronary arterial bypass graft or angioplasty; v) severe pulmonary, renal, or liver disease; vi) active substance abuse with alcohol or drugs by self-report; vii) active tobacco use (>8 cigarettes/day); viii) excessive alcohol consumption (>14 drinks per week for women or 21 drinks per week for men); ix) treatment with non-diabetes medications (e.g., corticosteroids, anti-psychotics) known to have metabolic/body weight effects that could affect the outcome measures or increase the risk of study procedures; x) history of bariatric surgery; xi) poorly controlled hypertension (SBP ≥160 mmHg or DBP ≥110 mmHg); xii) structured exercise >120 minutes/week; xiii) pregnant, lactating, not using effective birth control if premenopausal, or planning to become pregnant within the 12-month study period; xiv) unstable weight (>4% change in the last 2 months); xv) anemia (hemoglobin <10 g/dL); xvi) has a continuous glucose monitor (CGM) or plans to have a CGM in the next 12 months; xvii) major psychiatric illness that would interefer with study participation; and xviii) any person that is unable to provide informed consent or unwilling to complete the study or who, for any reason, the research team considers an inappropriate candidate for the study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline HbA1c to 6 months | Baseline and at the end of the intervention, at month 6
  To assess glycemic control

SECONDARY OUTCOMES:
Change from Baseline Insulin Sensitivity to 6 months | Baseline and end of the intervention, at month 6
  Insulin sensitivity assessed as HOMA-IR. The higher the score the more likely to be insulin resistant (less than 1.0 means insulin sensitivity, above 1.9 indicates early insulin resistance, above 2.9 indicates significant insulin resistance.
Change from Baseline Fasting Glucose to 6 months | Baseline and end of the intervention, at month 6
  Fasting glucose for those with T2D is below 131 mg/dL is optimal.
Change from Baseline Plasma Triglycerides to 6 months | Baseline and end of the intervention, at month 6
  Normal - Less than 150 milligrams per deciliter (mg/dL), or less than 1.7 millimoles per liter (mmol/L) Borderline high - 150 to 199 mg/dL (1.8 to 2.2 mmol/L) High - 200 to 499 mg/dL (2.3 to 5.6 mmol/L) Very high - 500 mg/dL or above (5.7 mmol/L or above)
Change from Baseline Systolic and Diastolic Blood Pressure to 12 months | Baseline and end of the intervention, at month 6
  To assess blood pressure changes. Normal is systolic: less than 120 mm Hg and diastolic: less than 80 mm Hg; At Risk (prehypertension) is systolic: 120-139 mm Hg and diastolic: 80-89 mm Hg; High Blood Pressure (hypertension) issystolic: 140 mm Hg or higher and diastolic: 90 mm Hg or higher
Change from Baseline Depressive Symptoms to 6 months | Baseline and end of the intervention, at month 6
  Depressive symptoms assessed by using the Patient Health Questionaire-9 (PHQ-9). The scale is from 0 to 27 with a higher score indicating worse depressive symptoms.
Change from Baseline Perceived Stress to 6 months | Baseline and end of the intervention, at month 6
  Stress assessed by using Perceived Stress Scale (PSS-4). The scale is from 0 to 16 with a higher score indicating more stress.
Change from Baseline Quality of Life to 6 months | Baseline and end of the intervention, at month 6
  Quality of life assessed by using the Health Survey Short Form (SF-12).Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

OTHER OUTCOMES:
Intervention Implementation Fidelity | During and at the end of the intervention, day 1 to day 183
  Fidelity to the delivery of the intervention will be quantified from a checklist of objectives the CHWs completes for each visit. The specific measure (e.g., the percent of content that was covered) will be verified by listening to audiotapes. The outcome variables for the participants include the participation in >80% of the sessions and the CHWs will note attendance of all participants in the study.
Intervention Implementation Acceptability | During and at the end of the intervention, day 1 to day 183
  Acceptability will be assessed using a newly formed 10-item questionnaire specific to the intervention for community health workers. For participants, a curated self-reported satisfaction survey will be developed.
Intervention Implementation Feasibility | During and at the end of the intervention, day 1 to day 183
  Feasibility will be assessed using a newly formed 10-item questionnaire specific to the intervention for community health workers. For participants, a curated self-reported satisfaction survey will be developed.
Intervention Implementation Adaptability | During and at the end of the intervention, day 1 to day 183
  Adaptability will be assessed by the community health workers annotating changes in their delivery of the intervention at every session.

CONTACTS AND LOCATIONS:
Overall Officials: Julia López, PhD, LCSW, Principal Investigator — Washington University School of Medicine
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez JE, Campbell KM. Racial and Ethnic Disparities in Prevalence and Care of Patients With Type 2 Diabetes. Clin Diabetes. 2017 Jan;35(1):66-70. doi: 10.2337/cd15-0048. No abstract available. PMID 28144049
- [Background] Aguayo-Mazzucato C, Diaque P, Hernandez S, Rosas S, Kostic A, Caballero AE. Understanding the growing epidemic of type 2 diabetes in the Hispanic population living in the United States. Diabetes Metab Res Rev. 2019 Feb;35(2):e3097. doi: 10.1002/dmrr.3097. Epub 2018 Dec 4. PMID 30445663
- [Background] Stacciarini JM, Shattell MM, Coady M, Wiens B. Review: Community-based participatory research approach to address mental health in minority populations. Community Ment Health J. 2011 Oct;47(5):489-97. doi: 10.1007/s10597-010-9319-z. Epub 2010 May 13. PMID 20464489
- [Background] Shah M, Kaselitz E, Heisler M. The role of community health workers in diabetes: update on current literature. Curr Diab Rep. 2013 Apr;13(2):163-71. doi: 10.1007/s11892-012-0359-3. PMID 23345198
- [Background] Yang X, Li Z, Sun J. Effects of Cognitive Behavioral Therapy-Based Intervention on Improving Glycaemic, Psychological, and Physiological Outcomes in Adult Patients With Diabetes Mellitus: A Meta-Analysis of Randomized Controlled Trials. Front Psychiatry. 2020 Jul 28;11:711. doi: 10.3389/fpsyt.2020.00711. eCollection 2020. PMID 32848906
- [Background] Walker RJ, Strom Williams J, Egede LE. Influence of Race, Ethnicity and Social Determinants of Health on Diabetes Outcomes. Am J Med Sci. 2016 Apr;351(4):366-73. doi: 10.1016/j.amjms.2016.01.008. PMID 27079342
- [Background] Schwab T, Meyer J, Merrell R. Measuring attitudes and health beliefs among Mexican Americans with diabetes. Diabetes Educ. 1994 May-Jun;20(3):221-7. doi: 10.1177/014572179402000308. PMID 7851237
- [Background] Fain JA. The Diabetes Educator (TDE): Successes, Opportunities, and Future Changes. Diabetes Educ. 2020 Dec;46(6):512-513. doi: 10.1177/0145721720976349. No abstract available. PMID 33353512
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Sep 10;140(11):e596-e646. doi: 10.1161/CIR.0000000000000678. Epub 2019 Mar 17. No abstract available. PMID 30879355